CLINICAL TRIAL: NCT03127358
Title: Smartphone Based Automated-Directly Observed Treatment Improves Adherence and SVR to Fixed-Dose Elbasvir and Grazoprevir in PWIDs: A Randomized Control Trial
Brief Title: Smartphone Based aDOT Treatment With Fixed-Dose Elbasvir and Grazoprevir in PWIDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: AiCure (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Julia H. Arnsten, Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-7215
Record Dates: First submitted 2017-03-24; First posted 2017-04-25 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis C; Medication Adherence
Keywords: Addiction; Sustained Viral Response; Adherence; Adverse Effects; Direct Acting Antiviral Agent; Chronic Hepatitis C; Resistance Development; Methadone Clinic; Primary Care; Directly Observed Therapy; Randomized Controlled Trial; Resistance; Reinfection; Treatment Outcome; Patient Navigation; Multi-Site; Liver Disease; Intervention
MeSH Terms: conditions — Hepatitis C; Medication Adherence; Behavior, Addictive; Hepatitis C, Chronic; Directly Observed Therapy; Reinfection; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- AiCure App (Experimental): Participants will use a-DOT technology called AiCure (a Smartphone App) to track ingestion of fixed-dose Elbasvir and Grazoprevir, 1 tablet, 50mg-100mg of each drug, respectively, daily for 12 weeks.
  Interventions: Device: AiCure
- Treatment As Usual (No Intervention): Participants will receive treatment for ingestion of fixed-dose Elbasvir and Grazoprevir, 1 tablet, 50mg-100mg of each drug, respectively, daily for 12 weeks without using the AiCure app.
- AiCure with gamification (Active Comparator): Sub-group of participants will use a-DOT technology called AiCure (a Smartphone app) with gaming to track ingestion of fixed-dose Elbasvir and Grazoprevir, 1 tablet, 50mg-100mg of each drug, respectively, daily for 12 weeks. The gaming feature is to test whether competition encourages engagement and helps to increase adherence to the HCV medication.
  Interventions: Device: AiCure with gamification

INTERVENTIONS:
Device: AiCure — Smartphone App
  Other Names: a-DOT, Smartphone App
  Arms: AiCure App
Device: AiCure with gamification — Smartphone App with gaming.
  Other Names: a-DOT with gamification
  Arms: AiCure with gamification

SUMMARY:
People who Inject Drugs (PWIDs) constitute 60% of the approximately 5 million people in the United States infected with hepatitis C virus (HCV). Successful HCV treatment leading to sustained viral response (SVR) is associated with increased survival, but to date successful treatment of PWIDs has been limited. Treatment of PWIDs is complex due to addiction, mental illness, poverty, homelessness, lack of positive social support, poor adherence-related skills, low motivation and knowledge, and poor access to and trust in the health care system. At Albert Einstein College of Medicine, the investigators have developed a multidisciplinary model of HCV care that integrates on-site primary care, substance abuse treatment, and HCV-related care within opiate agonist treatment clinics. To optimize HCV treatment outcomes, the investigators have introduced directly observed therapy (DOT). In the DOT model, one daily dose of oral HCV medication is administered with methadone. However, DOT is not feasible for PWIDs who are not enrolled in methadone maintenance treatment programs, and is less effective for methadone-maintained PWIDs who do not attend the methadone clinics every day. In addition, DOT has been used for decades both to measure and maximize adherence for treatment of tuberculosis infection, but the cost and logistical complexity of administering DOT for large HCV clinical programs would be prohibitive.

DETAILED DESCRIPTION:
Automated DOT (a-DOT), a smartphone app that uses facial recognition software and advanced features to detect non-ingestion, combines the accuracy of in-person DOT with the convenience of real-time centralized data collection and monitoring. Adding a daily side effect diary to a-DOT will further allow precise tracking of timing of both medication ingestion and side effects which may be compromising adherence. Zepatier (elbasvir and grazoprevir) is a new once-daily fixe-dose combination tablet which has achieved high rates of SVR ranging from 94 to 97 percent in genotype-1 infected patients including those with HIV/HCV coinfection and renal impairment. Zepatier is administered for 12 to 16 weeks, depending on HCV genotype, prior treatment history, and the presence of certain baseline NS5A polymorphisms (1a only). By administering Zepatier via this innovative a-DOT platform, the investigators hypothesize that PWIDs treated in real-wrold settings can be successfully treated with high rates of adherence and SVR.

In this proposed 18-month trials, 75 PWIDs enrolled in opiate agonist treatment (genotypes 1a and 1b) with chronic HCV will be enrolled over a 12-month period, and randomized to either aDOT or treatment as usual (TAU). The investigators will recruit PWIDs from diverse community settings include a syringe exchange program (NYHRE), federally-qualified health center (Comprehensive Health Care Center), homeless shelter (The Living Room), and a methadone maintenance treatment program (Montefiore Wellness Centers). All patients (inlcuding treatment-experienced and HIVV/HCV coinfected subjects) will be treated with Zepatier-based regimens as per the standard of care. Rigorous data are necessary to judge the contribution of a-DOT to the success of HCV treatment in PWIDs. By performing a randomized trial of a-DOT HCV therapy (Zepatier with and without ribavirin), the investigators will evaluate the efficacy of a-DOT for improving HCV treatment outcomes among PWIDs.

ELIGIBILITY:
Inclusion Criteria:

* HCV-infected (HCV RNA test above the limit of quantification at baseline)
* Genotypes/Subtypes: G1a or G1b
* Eligible for HCV treatment per 2016 AASLD/IDSA guidelines
* Willing to receive HCV treatment on-site at DoSA clinics
* Health care provider decision to treat patient with Zepatier-based therapy with or without ribavirin based on 2016 AASLD/IDSA guidelines
* Using illicit drugs (either opiates, cocaine, or benzodizepenes) within the last 6 months
* Age 18 or older
* Able to provide informed consent
* English or Spanish speaking

Exclusion Criteria:

* Known hypersensitivity (allergy) to elbasvir, grazoprevir, or ribavirin
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Arnsten, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Albert Einstein College of Medicine Division of Substance Abuse clinics, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates were from 11/14/17 to 7/20/18, during which 11 participants were recruited and enrolled into the study.
  Participants were recruited from a Montefiore Medical Center opioid treatment program in the Bronx. Participants were identified through chart review and provider referral, and through participant self-referral.
Period: Overall Study
Arm/Group | AiCure App | Treatment As Usual | AiCure With Gamification
Started | 3 (3/9/18:Date first participant was randomized to this arm.) | 3 (3/22/18: Date first participant randomized to this arm.) | 5 (3/14/18: Date first participant randomized to this arm..)
Completed | 3 (12/26/18: Date of SVR for last participant randomized to this arm.) | 3 (2/6/19: Date of SVR for last participant randomized to this arm.) | 5 (11/20/18: Date of SVR for last participant randomized to this arm.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AiCure App: Direct Observed Therapy via the AiCure app (a-DOT)
- Total: Total of all reporting groups
Arm/Group | AiCure App | Treatment As Usual | AiCure With Gamification | Total
Number analyzed (Participants) | 3 | 3 | 5 | 11
Age, Continuous [Mean (Full Range); unit: years] | 53 [43 to 59] | 60 [40 to 71] | 58 [50 to 66] | 57 [43 to 71]
Sex: Female, Male [Count of Participants; unit: Participants] — Select one of the following:
  Male, Female, other (describe)
  Participants
    Female | 1 | 0 | 2 | 3
    Male | 2 | 3 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — count of participants who identified their ethnicity as Hispanic/Latino
  Participants
    Hispanic or Latino | 1 | 1 | 4 | 6
    Not Hispanic or Latino | 2 | 2 | 1 | 5
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 4
  White | 0 | 2 | 4 | 6
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: HCV Treatment Adherence
Description: The amount of medication taken by each patient during the treatment period is expressed as a percentage (range 0-100%). Subjects will be classified as "adherent" if they receive at least 80% of the total dose of Zepatier. The numbers below denotes the mean percent of the medication the participants in each arm took.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: percent of medication taken
Arm/Group | AiCure App | Treatment As Usual | AiCure With Gamification
Number analyzed (Participants) | 3 | 3 | 5
percent of medication taken | 83 [0 to 100] | 100 [0 to 100] | 88 [0 to 100]

2. Secondary Outcome: Number of Participants With HCV Treatment Completion
Description: Participants will be considered to have completed treatment if they have completed at least 80% of the planned treatment course (e.g. at least 10 week of 12-week course).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- AiCure App: Participants will use a-DOT technology called AiCure (a Smartphone App) to track ingestion of fixed-dose Elbasvir and Grazoprevir, 1 tablet, 50mg-100mg of each drug, respectively, daily for 12 weeks.
  AiCure: Smartphone App
  3 out 3 patients completed HCV treatment.
- Treatment As Usual: Participants will receive treatment for ingestion of fixed-dose Elbasvir and Grazoprevir, 1 tablet, 50mg-100mg of each drug, respectively, daily for 12 weeks without using the AiCure app.
  3 out 3 patients completed HCV treatment.
- AiCure With Gamification: Sub-group of participants will use a-DOT technology called AiCure (a Smartphone app) with gaming to track ingestion of fixed-dose Elbasvir and Grazoprevir, 1 tablet, 50mg-100mg of each drug, respectively, daily for 12 weeks. The gaming feature is to test whether competition encourages engagement and helps to increase adherence to the HCV medication.
  AiCure with gamification: Smartphone App with gaming.
  5 out 5 patients completed HCV treatment.
Arm/Group | AiCure App | Treatment As Usual | AiCure With Gamification
Number analyzed (Participants) | 3 | 3 | 5
Participants | 3 | 3 | 5

3. Secondary Outcome: Number of Participants With Sustained Viral Response (SVR)
Description: HCV viral load undectable 12 weeks after treatment completion. Undetectable HCV viral load is defined as <15 IU/ml and "target not detected". IU refers to "international units".One of the main outcomes looked for was the amount of patients who achieved Sustained Virologic Response (SVR) at 12 weeks post treatment, which denotes a cure of Hepatitis C.
Time Frame: 12 weeks post treatment
Measure: Number; unit: percent of patients with SVR
Groups:
- AiCure App: Participants will use a-DOT technology called AiCure (a Smartphone App) to track ingestion of fixed-dose Elbasvir and Grazoprevir, 1 tablet, 50mg-100mg of each drug, respectively, daily for 12 weeks.
  AiCure: Smartphone App
  3 out 3 patients achieved SVR.
- Treatment As Usual: Participants will receive treatment for ingestion of fixed-dose Elbasvir and Grazoprevir, 1 tablet, 50mg-100mg of each drug, respectively, daily for 12 weeks without using the AiCure app.
  3 out 3 patients achieved SVR.
- AiCure With Gamification: Sub-group of participants will use a-DOT technology called AiCure (a Smartphone app) with gaming to track ingestion of fixed-dose Elbasvir and Grazoprevir, 1 tablet, 50mg-100mg of each drug, respectively, daily for 12 weeks. The gaming feature is to test whether competition encourages engagement and helps to increase adherence to the HCV medication.
  AiCure with gamification: Smartphone App with gaming.
  5 out 5 patients achieved SVR.
Arm/Group | AiCure App | Treatment As Usual | AiCure With Gamification
Number analyzed (Participants) | 3 | 3 | 5
percent of patients with SVR | 100 | 100 | 100

ADVERSE EVENTS:
Time Frame: The study participants were assessed from 4 months prior to enrollment, through 12 weeks of treatment, to 7 months after treatment, an average of 14 months
Description: The definition of adverse event and/or serious adverse event does not differ from the definitions on clinicaltrials.gov.
Arm/Group | AiCure App | Treatment As Usual | AiCure With Gamification
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5

LIMITATIONS AND CAVEATS:
Early termination due to discontinued funding led to small numbers of subjects analyzed, and study personnel were no longer available to work on this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT03127358/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT03127358/ICF_001.pdf